CLINICAL TRIAL: NCT04677439
Title: Efficacy and the Safety of Flumatinib in Treatment of CML-CP Patients With Ph+ Post Imatinib Failure
Brief Title: Flumatinib in CML-CP Patients With Ph+ Post Imatinib Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: Hainan General Hospital (Other); Sanya Central Hospital (Unknown); First Affiliated Hospital of Shantou University Medical College (Other); Peking University Shenzhen Hospital (Other); Dongguan People's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Flumatinib20201216
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Flumatinib; Chronic Myeloid Leukemia, Chronic Phase; Imatinib
Keywords: Flumatinib, CML-CP with Ph+
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — flumatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flumatinib (Experimental)
  Interventions: Drug: Flumatinib

INTERVENTIONS:
Drug: Flumatinib — 600 mg of Flumatinib orally daily for 24 months

SUMMARY:
The purpose of this study is to explore the efficacy and safety of flumatinib in chronic phase of chronic myeloid leukemia (CML-CP) patients With Ph+ post imatinib failure.

DETAILED DESCRIPTION:
A multicenter, single-arm, prospective, open-label study to detect the efficacy and safety of flumatinib by measuring rates of major molecular response (MMR) at 12 months in CML-CP patients with Ph+ in China. Approximately 200 Patients will be recruited consecutively from the study sites during the enrollment period and will be given flumatinib 600 mg QD. The duration of patient participation will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of CML-CP with Ph+.
* ECOG performance of 0-2.
* Adequate end organ function defined as the following: total bilirubin <1.5x ULN, SGPT <2.5x ULN, creatinine <1.5x ULN.
* Treatment failure after imatinib at 3 or 6 months with BCR-ABL >10%.
* Patients must sign an informed consent form (ICF) indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.

Exclusion Criteria:

* Previously documented T315I mutation.
* History of TKI treatments except of imatinib.
* History of undergone major surgery within 4 weeks.
* Patients unwilling or unable to comply with the protocol.
* Pregnant or breast-feeding patients.
* patients with other malignant tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve and maintain MMR at 12 months using RQ-PCR test. | 12 months
  Major molecular response (MMR) is defined as BCR-ABL1 ≤ 0.1 percent.

SECONDARY OUTCOMES:
Proportion of patients with MR 4.0 at 3, 6, 9, 12 months. | 3, 6, 9, 12 months.
  Molecular response (MR) 4.0 is defined as BCR-ABL transcripts ≤ 0.01 percent.
Proportion of patients with MR 4.5 at 3, 6, 9, 12 months. | 3, 6, 9, 12 months.
  Molecular response (MR) 4.5 is defined as BCR-ABL transcripts ≤ 0.0032 percent.
Proportion of patients with MMR at 3, 6, 9 months. | 3, 6, 9 months
Incidence of adverse events (AEs) and serious adverse events (SAEs) to Flumatinib. | 24 months
  Evaluation of adverse events (AEs), serious AEs (SAEs), and clinically relevant changes in laboratory tests according to laboratory reference ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Du, Phd, Principal Investigator — Shenzhen Second People's Hospital
Locations (1):
- The Second People's Hospital of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No